CLINICAL TRIAL: NCT03308838
Title: A Case-control Study of Costa Rican Adults With Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Universidad de Costa Rica (Other); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Ana Baylin, Associate Professor, University of Michigan
Other Study IDs: HUM00037337
Record Dates: First submitted 2017-10-09; First posted 2017-10-13 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Myocardial Infarction, Acute
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — We collected adipose tissue biopsies to quantify adipose tissue fatty acids.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Cases consisted of Costa Rican adults who were diagnosed as survivors of a first acute myocardial infarction.
- Controls: Controls consisted of healthy individuals randomly identified from the underlying source population in Costa Rica and matched to each case by age, sex, and area of residence.

SUMMARY:
This observational case-control trial sought to identify and characterize different exposures associated with nonfatal acute myocardial infarction in Costa Rican adults. Exposures assessed included dietary variables and adipose tissue fatty acids.

ELIGIBILITY:
Inclusion Criteria:

* Cases were eligible if they met the World Health Organization criteria for MI

Exclusion Criteria (Cases):

* Died during hospitalization
* Were 75 years or older on the day of their first MI
* Were physically or mentally unable to answer the questionnaire
* Had a previous hospital admission related to cardiovascular disease

Exclusion Criteria (Controls):

* Ever had an MI
* Were physically or mentally unable to answer the questionnaire

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Cases were survivors of a first acute MI as diagnosed by a cardiologist at any of the six recruiting hospitals in the Central Valley of Costa Rica. Controls were population-based controls from Costa Rica.
Sampling Method: Probability Sample
Enrollment: 4547 (Actual)
Dates: Start 1994-08-01 (Actual); Primary Completion 2004-08-01 (Actual); Study Completion 2004-08-01 (Actual)

PRIMARY OUTCOMES:
Nonfatal Acute Myocardial Infarction | 1994-2004
  Identified by independent examinations of two cardiologists at any of the six recruiting hospitals in the catchment area of the Central Valley of Costa Rica. Outcome was determined as being met if they met the World Health Organization criteria for myocardial infarction.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Baylin, MD, DrPH, Principal Investigator — University of Michigan
Locations (1):
- University of Costa Rica, San Pedro, Provincia de San José, Costa Rica

IPD SHARING:
Plan to Share IPD: No
The data are completely de-identified.

REFERENCES:
- [Result] El-Sohemy A, Baylin A, Spiegelman D, Ascherio A, Campos H. Dietary and adipose tissue gamma-tocopherol and risk of myocardial infarction. Epidemiology. 2002 Mar;13(2):216-23. doi: 10.1097/00001648-200203000-00018. PMID 11880764
- [Result] Baylin A, Kabagambe EK, Ascherio A, Spiegelman D, Campos H. Adipose tissue alpha-linolenic acid and nonfatal acute myocardial infarction in Costa Rica. Circulation. 2003 Apr 1;107(12):1586-91. doi: 10.1161/01.CIR.0000058165.81208.C6. Epub 2003 Mar 10. PMID 12668490
- [Result] Baylin A, Kabagambe EK, Ascherio A, Spiegelman D, Campos H. High 18:2 trans-fatty acids in adipose tissue are associated with increased risk of nonfatal acute myocardial infarction in costa rican adults. J Nutr. 2003 Apr;133(4):1186-91. doi: 10.1093/jn/133.4.1186. PMID 12672941
- [Result] Kabagambe EK, Baylin A, Campos H. Nonfatal acute myocardial infarction in Costa Rica: modifiable risk factors, population-attributable risks, and adherence to dietary guidelines. Circulation. 2007 Mar 6;115(9):1075-81. doi: 10.1161/CIRCULATIONAHA.106.643544. PMID 17339565
- [Result] Aslibekyan S, Campos H, Loucks EB, Linkletter CD, Ordovas JM, Baylin A. Development of a cardiovascular risk score for use in low- and middle-income countries. J Nutr. 2011 Jul;141(7):1375-80. doi: 10.3945/jn.110.133140. Epub 2011 May 11. PMID 21562240
- [Result] Wang D, Campos H, Baylin A. Red meat intake is positively associated with non-fatal acute myocardial infarction in the Costa Rica Heart Study. Br J Nutr. 2017 Aug;118(4):303-311. doi: 10.1017/S000711451700201X. PMID 28875869